CLINICAL TRIAL: NCT00723281
Title: Comparison of CT Angiography With Conventional Angiography and Intravascular Ultrasound in Heart Transplant Patients
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: American Roentgen Ray Society (Other)
Responsible Party: Principal Investigator, Karen Ordovas, Assistant Professor, University of California, San Francisco
Other Study IDs: H627-29905
Record Dates: First submitted 2008-07-24; First posted 2008-07-28 (Estimated); Last update posted 2019-06-17 (Actual); Status verified 2019-06

CONDITIONS: Heart Transplantation; Coronary Artery Disease
Keywords: transplant coronary artery disease; CT angiography; conventional angiography; intravascular ultrasound; Heart transplant patients with known transplant coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The overall goal of this study is to determine if non-invasive imaging with state of the art CT coronary angiography can be used to screen for transplant coronary artery disease in the setting of heart transplant.

Our current protocol at UCSF for heart transplant patients involves screening with stress tests as well as coronary angiograms with intravascular ultrasound to assess the diameter of the lumen of the coronary arteries and to assess wall thickness.

DETAILED DESCRIPTION:
Our hypothesis is that state of the art CT coronary angiography can be used to acquire data regarding the coronary arteries in the setting of heart transplant and be used to risk stratify patients with regards to the developments of transplant coronary artery disease.

Specific Aim 1- To test the hypothesis that coronary CTA can accurately measure cross-sectional vessel wall area using conventional coronary angiography with intra-vascular ultrasound as the standard of reference.

Specific Aim 2- To test the hypothesis that coronary CTA can accurately measure cross-sectional vessel wall thickness, vessel area and luminal area using conventional coronary angiography with intra-vascular ultrasound as the standard of reference.

Secondary Aim - To asses the correlation of cross-sectional vessel wall area, vessel wall thickness, vessel area, luminal area and vessel wall index with global and regional left ventricular function using coronary CTA.

ELIGIBILITY:
Inclusion Criteria:

1. Patient referred for coronary angiography and IVUS as part of their standard clinical care;
2. Patients must be 18 years of age or older.
3. Any ethnic background is acceptable.

Exclusion Criteria:

1. Patients with contraindications for the use of iodinated contrast (allergic reaction, renal failure, multiple myeloma, etc) will be excluded.
2. Patients with heart rate higher than 65 bpm and contraindications for the use of beta-blockers, listed below:

   Systolic blood pressure < 90mmHg Decompensated congestive heart failure; COPD or asthma in use of bronchodilator; Second or third degree heart block; Severe aortic stenosis, defined by a pressure gradient higher than 50 mmHg and/or the presence of symptoms.
3. Patients with contraindications for the use of nitroglycerin, listed below:

   Severe anemia; Increased intracranial pressure; Known hypersensitivity; Use of Sildenafil Citrate (Viagra®)
4. Children and pregnant women will be excluded because of risks associated with radiation exposure.
5. Patients must have no atrial fibrillation, as this will interfere with cardiac gating for the examination.
6. Patients unable to give informed consent will be excluded as well.
7. Patients with a coronary stent placed.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All heart transplant patients at UCSF with known transplant coronary artery disease will be candidates for the study
Sampling Method: Non-Probability Sample
Enrollment: 18 (Estimated)
Dates: Start 2007-01; Primary Completion 2010-07 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Based on these considerations, 18 patients will be recruited to participate in this study, including at least 10 patients with coronary allograft vasculopathy. Only CTA of patients with positive echocardiographic stress test will be included in the study | CTA studies will be done in an interval of 1 day to 30 days before the invasive studies

CONTACTS AND LOCATIONS:
Overall Officials: Charles B Higgins, MD, Principal Investigator — UCSF Department of Radiology
Locations (1):
- UCSF Medical Center, San Francisco, California, United States

REFERENCES:
- [Background] Mehra MR, Ventura HO, Chambers R, Collins TJ, Ramee SR, Kates MA, Smart FW, Stapleton DD. Predictive model to assess risk for cardiac allograft vasculopathy: an intravascular ultrasound study. J Am Coll Cardiol. 1995 Nov 15;26(6):1537-44. doi: 10.1016/0735-1097(95)00357-6. PMID 7594082
- [Background] Zakliczynski M, Swierad M, Zakliczynska H, Maruszewski M, Buszman P, Zembala M. Usefulness of stanford scale of intimal hyperplasia assessed by intravascular ultrasound to predict time of onset and severity of cardiac allograft vasculopathy. Transplant Proc. 2005 Mar;37(2):1343-5. doi: 10.1016/j.transproceed.2004.12.143. PMID 15848715
- [Background] Leber AW, Becker A, Knez A, von Ziegler F, Sirol M, Nikolaou K, Ohnesorge B, Fayad ZA, Becker CR, Reiser M, Steinbeck G, Boekstegers P. Accuracy of 64-slice computed tomography to classify and quantify plaque volumes in the proximal coronary system: a comparative study using intravascular ultrasound. J Am Coll Cardiol. 2006 Feb 7;47(3):672-7. doi: 10.1016/j.jacc.2005.10.058. Epub 2006 Jan 6. PMID 16458154
- [Background] Moselewski F, Ropers D, Pohle K, Hoffmann U, Ferencik M, Chan RC, Cury RC, Abbara S, Jang IK, Brady TJ, Daniel WG, Achenbach S. Comparison of measurement of cross-sectional coronary atherosclerotic plaque and vessel areas by 16-slice multidetector computed tomography versus intravascular ultrasound. Am J Cardiol. 2004 Nov 15;94(10):1294-7. doi: 10.1016/j.amjcard.2004.07.117. PMID 15541250
- [Background] Sigurdsson G, Carrascosa P, Yamani MH, Greenberg NL, Perrone S, Lev G, Desai MY, Garcia MJ. Detection of transplant coronary artery disease using multidetector computed tomography with adaptative multisegment reconstruction. J Am Coll Cardiol. 2006 Aug 15;48(4):772-8. doi: 10.1016/j.jacc.2006.04.082. Epub 2006 Jul 25. PMID 16904548
- [Background] Gregory SA, Ferencik M, Achenbach S, Yeh RW, Hoffmann U, Inglessis I, Cury RC, Nieman K, McNulty IA, Laffan JA, Pomerantsev EV, Brady TJ, Semigran MJ, Jang IK. Comparison of sixty-four-slice multidetector computed tomographic coronary angiography to coronary angiography with intravascular ultrasound for the detection of transplant vasculopathy. Am J Cardiol. 2006 Oct 1;98(7):877-84. doi: 10.1016/j.amjcard.2006.04.027. Epub 2006 Aug 4. PMID 16996866
- [Background] Ferencik M, Moselewski F, Ropers D, Hoffmann U, Baum U, Anders K, Pomerantsev EV, Abbara S, Brady TJ, Achenbach S. Quantitative parameters of image quality in multidetector spiral computed tomographic coronary imaging with submillimeter collimation. Am J Cardiol. 2003 Dec 1;92(11):1257-62. doi: 10.1016/j.amjcard.2003.08.003. PMID 14636899
- [Background] Obuchowski NA. Estimating and comparing diagnostic tests' accuracy when the gold standard is not binary. Acad Radiol. 2005 Sep;12(9):1198-204. doi: 10.1016/j.acra.2005.05.013. PMID 16099683
- [Background] Obuchowski NA. An ROC-type measure of diagnostic accuracy when the gold standard is continuous-scale. Stat Med. 2006 Feb 15;25(3):481-93. doi: 10.1002/sim.2228. PMID 16287217
- [Background] Efron B, Tibshirani R. An Introduction to the Bootstrap. New York: Chapman and Hall; 1993
- [Background] Kish. Survey Sampling. New York: Wiley & Sons; 1965.
- [Background] Lachin JM. Introduction to sample size determination and power analysis for clinical trials. Control Clin Trials. 1981 Jun;2(2):93-113. doi: 10.1016/0197-2456(81)90001-5. PMID 7273794
- [Background] Pannu HK, Alvarez W Jr, Fishman EK. Beta-blockers for cardiac CT: a primer for the radiologist. AJR Am J Roentgenol. 2006 Jun;186(6 Suppl 2):S341-5. doi: 10.2214/AJR.04.1944. PMID 16714607